CLINICAL TRIAL: NCT06157632
Title: Role of Preoperative Serum Thyroglobulin Level to Differentiate Between Different Thyroid Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Hussein Hasan, Resident doctor at general surgery departement assiut university, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Thyroglobulin level
Record Dates: First submitted 2023-11-15; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Level of Thyrogobulin in Different Thyroid Nodules

STUDY DESIGN:
Intervention Model Description: patients with thyoid nodules that will do thyriodectomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with thyoid nodules (Other): Patients with thyroid nodules that will do thyroidectomy
  Interventions: Procedure: Thyriodectomy

INTERVENTIONS:
Procedure: Thyriodectomy — Thyroidectomy

SUMMARY:
Role of preoperative serum thyroglobulin level to differentiate between different thyroid nodules

DETAILED DESCRIPTION:
Incidence of thyroid nodules varies according to the methods of diagnosis, 4-7% by palpation and 17-67% by high resolution ultrasound.

The gold standard of diagnosis for thyroid nodules is fine needle aspiration (FNA); however, fine needle aspiration cytology (FNAC) alone is insufficient to detect cancer because of inadequate cytology (5-15%) and in cases of follicular neoplasm (15-25%) where only surgery is diagnostically conclusive. Therefore, other factors in addition to FNA should be considered to predict malignancy. This study is done to evaluate the association between elevated pre-operative thyroglobulin levels and histopathologically proven thyroid carcinoma.

Metabolism of thyroglobulin occurs in the liver and via thyroid gland and recycling of the protein takes place. Circulating thyroglobulin features a half lifetime of 65 hours. Following thyroidectomy, it will take many weeks before thyroglobulin levels become undetectable. After thyroglobulin levels become undetectable (following thyroidectomy), levels are often serially monitored.

A subsequent elevation of the thyroglobulin level is an indicator of recurrence of papillary or follicular thyroid carcinoma. Hence, thyroglobulin levels in the blood are mainly used as a tumor marker for certain kinds of thyroid cancer (particularly papillary or follicular thyroid cancer). Thyroglobulin is not produced by medullary or anaplastic carcinoma.

Therefore, this study tries to evaluate the association between the preoperative thyroglobulin levels and thyroid carcinoma proven by post-operative histopathology.

ELIGIBILITY:
Inclusion Criteria:

1. age between 15 to 70 years old
2. patients with solitary thyroid nodules
3. pateints who are fit for surgeries

Exclusion Criteria:

* 1_patients who are unfit for surgeries

  2_ age below 15 years and above 70 years old

  3-patients with thyroid nodule receiving drugs that affect thyroglobulin level as iodine

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patients with thyroid nodules
Enrollment: 30 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-11-18 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
Role of preoperative serum thyroglobulin level to differentiate between different thyroid nodules | Two year
  Use of serum thyroglobulin to differentiate between different thyroid nodules preoperoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Baker, Prof, Study Director — Assiut University; Mahmoud Thabet, Assistant.prof, Study Director — Assiut University